CLINICAL TRIAL: NCT05141461
Title: The Effect of Intravenous Dexamethasone on Rebound Pain After Interscalene Brachial Plexus Block for Shoulder Surgery: a Randomized Controlled Trial
Brief Title: The Effect of Intravenous Dexamethasone on Rebound Pain After Interscalene Brachial Plexus Block for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-2021/13
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2021-10

CONDITIONS: Rebound Pain
Keywords: interscalene brachial plexus block; shoulder surgery; dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study investigators will not be aware of what group the participant belongs to when assessing the patient at post-operative period
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Sham Comparator): The patients will be received an ultrasound-guided interscalene brachial plexus block with 15 mL bupivacaine 0.5%.
  Interventions: Procedure: Group C
- Group Dex (Experimental): The patients will be received an ultrasound-guided interscalene brachial plexus block with 15 mL bupivacaine 0.5% and 5 mg intravenous dexamethasone.
  Interventions: Procedure: Group Dex

INTERVENTIONS:
Procedure: Group C — Patients will receive 2 mg midazolam and 50 ug fentanyl for sedation before the block procedure. Each patient will be positioned appropriately, then a high-frequency linear array transducer (13-6 MHz) will be placed in the interscalene region to define the brachial plexus on the short axis. Under sterile conditions, a 50 mm block needle will be advanced into the interscalen area using the in-plane method. After localization and negative aspiration, 15 ML of 5% bupivacaine drug will be injected into the interscalene area. 100 ml of NACI will be given intravenously within 15 minutes.
  General anesthesia will be performed using 2 mg/kg of propofol and 1-2 µg/kg of fentanyl. Tracheal intubation will be facilitated with 0.6mg/kg rocuronium. Anesthesia will be maintained using 50% oxygen and 2% sevoflurane. Patients will be extubated into the operating room after reversing residual muscle relaxation. A multimodal analgesia regimen will be applied postoperatively.
  Arms: Group C
Procedure: Group Dex — Patients will receive 2 mg midazolam and 50 ug fentanyl for sedation before the block procedure. Each patient will be positioned appropriately, then a high-frequency linear array transducer (13-6 MHz) will be placed in the interscalene region to define the brachial plexus on the short axis. Under sterile conditions, a 50 mm block needle will be advanced into the interscalene area using the in-plane method. After localization and negative aspiration, 15 ML of 5% bupivacaine drug will be injected into the interscalene area. 5 mg dexamethasone intravenously will be given in 100 ml NACI within 15 minutes.
  General anesthesia will be performed using 2 mg/kg of propofol and 1-2 µg/kg of fentanyl. Tracheal intubation will be facilitated with 0.6mg/kg rocuronium. Anesthesia will be maintained using 50% oxygen and 2% sevoflurane. Patients will be extubated into the operating room after reversing residual muscle relaxation. A multimodal analgesia regimen will be applied postoperatively.
  Arms: Group Dex

SUMMARY:
The rebound pain after nerve block could interfere with the patient's recovery and rehabilitation. It is not known how intravenous dexamethasone affects rebound pain. This study aims to evaluate the effect of intravenous dexamethasone on rebound pain after interscalene block for shoulder surgery.

DETAILED DESCRIPTION:
Shoulder rotator cuff repair and acromioplasty are associated with severe postoperative pain. The interscalene block (ISB) is commonly used for this type of surgery, providing analgesia by anesthetizing the nerves that supply the shoulder. Although the nerve block provides extremely effective analgesia for the first 6-8 hours, patients experience severe pain once its effect has been wearing off. Rebound pain is a severe pain that occurs when the effect of a nerve block disappears in a patient during the postoperative period. The purpose of this study is to investigate whether the use of intravenous dexamethasone reduces rebound pain in patients recruiting for shoulder surgery with interscalene brachial plexus blockade.

This study will be conducted as a single-center, prospective, randomized, double-blinded trial in a university hospital. Patients scheduled for elective shoulder surgery will be screened for enrollment in the study. All subjects will undergo ultrasound-guided interscalene nerve block before induction of general anesthesia. They will be randomly assigned into the two groups which use intravenous dexamethasone or not. An anesthesiologist who will perform blocks will not involve in the data collection. Other health care workers who will involve in the evaluation of postoperative pain scores, nausea and vomiting, opioid consumption, quality of Sleep, and Quality of Recovery score will be blinded to the group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing shoulder surgery
* Having signed a written informed consent form,
* ASAI-III

Exclusion Criteria:

* Inadequate indication for interscalene block (Coagulation disorder, local infection of block site, Diaphragmatic paralysis, Allergy to local anesthetics)
* Neuropathic disorder
* Severe cardiopulmonary disease
* Systemic steroid use
* Chronic opioids use
* Stomach ulcer
* Ucontrolled Diabetes
* Psychiatric disorders,
* Pregnancy,
* Severe obesity (body mass index > 35 kg/m2)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
The difference of pain score before and after interscalene block resolution | First 12 hours after interscalene block effect disappears
  The difference in the pain score between when the block is working and when it has resolved. Pain scores (0 = no pain; 10 = worst pain imaginable) using a Numerical Rating Scale (NRS) ranging from 0 to 10.
Incidence of rebound pain | One week after surgery
  Rebound pain is described as severe pain (NRS ≥ 7)

SECONDARY OUTCOMES:
Analgesic consumption | Postoperative 48 hours
  Rescue analgesic consumption in the first 48 hours postoperatively will be recorded.
Quality of Recovery 15 Score | Postoperative day 1 and day 7
  Quality of Recovery (QoR)-15 survey.Minimum value: 0, Maximum value: 150, higher scores mean better.
Numeric Rating Scale pain score ( NRS) | Postoperative 48 hours
  Pain scores (0 = no pain; 10 = worst pain imaginable) using a Numerical Rating Scale (NRS) ranging from 0 to 10. It will be recorded at the 2nd, 4th, 6th, 8th, 12th, 16th, 18th, and 24th hours in the postoperative period
Interscalene block resolution time | Postoperative 24 hours
  The time of the first analgesic request. If the patient will not need analgesic, the block will be accepted as resolved when numbness or heaviness will not be felt by the patient.
Glucose measurement | Postoperative 24th hour
  Glucose measurement
Number of Participants with Surgical infection | Postoperative 14 days
  Number of Participants diagnosed with surgical infection
Sleep Quality measured with Likert Scale | One week after surgery
  Patients' perceived sleep quality will be assessed with a Likert scale. Likert scale is scored from Likert scale where 1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied and 5 = very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Başaran, MD,DESA, Study Director — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)